CLINICAL TRIAL: NCT01314508
Title: Increlex Treatment of Children With Chronic Liver Disease and Short Stature
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor has notified us that they are not funding the study
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Anna Haddal, M.D., UCLA Department of Pediatrics, Division of Pediatric Endocrinology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-03-018
Record Dates: First submitted 2011-03-08; First posted 2011-03-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Growth Failure; Chronic Liver Disease
Keywords: pre-pubertal children; pre-transplant; not treated with growth hormone for at least 3 months
MeSH Terms: conditions — Failure to Thrive | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients will be treated with IGF-1 factors (Other): Patients will serve as their own control.
  Interventions: Drug: Increlex

INTERVENTIONS:
Drug: Increlex — Increlex therapy will begin at 40 micrograms/kg/day twice a day. The dose will be escalated by 20 mcg twice a day every other week up to 100mcg/kg/week.

SUMMARY:
A major consequence of chronic liver disease in childhood is growth failure. This is because a chemical essential for growth called growth factor is created in the liver. Lack of response to growth hormone in people with chronic liver disease is characterized by high levels of growth hormone and low levels of growth factors. This growth hormone resistance is reflected in a variety of factors including insulin resistance and low nutritional intake. Unfortunately, growth hormone therapy has no effect for children with liver disease. In addition, failure of normal growth or malnutrition makes liver disease even worse in children, and growth hormone therapy is not likely to reverse this. A lack of proper nutrition is associated with hospitalizations and frequent complications. Poor growth is a predictor of poor outcomes after liver transplantation. Thus the management of children with liver disease remains a challenge. Children who have successful orthotopic liver transplants (OLT) show much improvement in some aspects of growth, including skin fold thickness, mid-arm circumference, and normalization of growth factor levels. However, some studies have recently reported that the growth of 15-20% of children remains poor even after a liver transplant. This can be explained by persistent abnormalities in growth factors after transplant.

Growth factor was found to be a good tool for prognosis in patients with chronic liver disease. Studies showed that patients with liver cirrhosis and growth factor levels below normal values showed lower long-term survival rates compared with patients who had above normal values. This suggests that growth factor can be a good predictor of survival and early marker of poor liver function. In this case, aggressive feeding may modestly improve growth factor levels leading to improved growth but it is unlikely that effects will be optimal. The investigators propose that growth factor administration may have a positive effect that leads to better growth which is a major predictor of good outcome. To date, no reports study the use of growth factor in children with chronic liver disease. This study proposes to examine the effect of growth factor therapy in childhood chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

Pre liver transplant patients with:

* Chronic liver disease
* Short stature (< 5%)
* Low IGF-1 (<-1SDS for age)
* Chronologic age 4-18 and bone age < 14 for boys and < 12 for girls (pre-pubertal)

Exclusion Criteria:

* Status post transplant
* Evidence of malignancy
* Diabetes mellitus
* Participation in other clinical trials involving investigational products
* Treatment with growth hormone within 3 months
* Pregnancy
* Significant abnormality in clinical results
* Hypoglycemic at baseline
* Allergic to benzyl alcohol

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Growth velocity is the primary outcome. Improved height SDS | One year of therapy
  Improved growth velocity with improved height standard deviation scores (SDS) is the primary expected result.

SECONDARY OUTCOMES:
Improved BMI | 12 months
  An improved body mass index is a secondary expected result of this study.
Improved quality of life | 12 months
  An improved quality of life as assessed by the Pediatric Quality of Life Inventory forms is another expected result.